CLINICAL TRIAL: NCT00619957
Title: Two-year Study to Determine the Efficacy and Safety of Risedronate Therapy Administered 35 mg Once A Week in Men With Osteoporosis for 2 Years Followed by a 2 Year Open Label Study
Brief Title: Efficacy and Safety of Risedronate Therapy Administered 35 mg Once A Week in Men With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001092 and 2001092 OL
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-09

CONDITIONS: Other Osteoporosis
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo tablet once a week for 2 years followed by once a week Risedronate for 2 years
  Interventions: Drug: Placebo tablet
- Risedronate (Experimental): 35 mg risedronate tablet once a week for 2 years followed by open label 35 mg risedronate once a week for 2 years
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Placebo tablet — one placebo once a week for two years followed by one 35 mg risedronate once a week for two years
  Arms: 1
Drug: Risedronate — one 35 mg risedronate once a week for two years followed by one 35 mg risedronate once a week for two years
  Arms: Risedronate

SUMMARY:
Two year study to determine the safety and efficacy of weekly 35 mg Risedronate doses in men with osteoporosis followed by a two year follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Documented osteoporosis of the femoral neck and lumbar spine

Exclusion Criteria:

* BMI greater than or equal to 35

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2002-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich Wenderoth, MD, Study Director — Procter and Gamble
Locations (23):
- United States (7):
  - Research Site, Palm Desert, California
  - Research Site, Lakewood, Colorado
  - Research Site, Stuart, Florida
  - Research Site, St Louis, Missouri
  - Research Facility, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Wyomissing, Pennsylvania
- Australia (2):
  - Research Facility, Concord
  - Research Facility, Heidelburg
- Research Facility, Leuven, Belgium
- Research Site, Prague, Czechia
- France (2):
  - Research Facility, Angers
  - Research Site, Lyon
- Hungary (2):
  - Research Facility, Budapest
  - Research Site, Budapest
- Research Site, Beirut, Lebanon
- Research Site, Rotterdam, Netherlands
- Poland (3):
  - Research Site, Bialystok
  - Research Site, Warsaw
  - Research Site, Wroclaw
- United Kingdom (3):
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Sheffield

REFERENCES:
- [Derived] Boonen S, Lorenc RS, Wenderoth D, Stoner KJ, Eusebio R, Orwoll ES. Evidence for safety and efficacy of risedronate in men with osteoporosis over 4 years of treatment: Results from the 2-year, open-label, extension study of a 2-year, randomized, double-blind, placebo-controlled study. Bone. 2012 Sep;51(3):383-8. doi: 10.1016/j.bone.2012.06.016. Epub 2012 Jun 30. PMID 22750403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 03 Jun 2002.
Groups:
- Placebo: Placebo tablet once a week for 2 years followed by once a week Risedronate 35 mg tablet for 2 years
- Risedronate: 35 mg risedronate tablet once a week for 2 years followed by an open label with 35 mg risedronate once a week for 2 years
Period: Month 24 Double-Blind
Arm/Group | Placebo | Risedronate
Started | 93 | 192
Intent to Treat (ITT Population) | 93 | 191 (One subject did not take any study medication.)
Completed | 75 | 175
Not Completed | 18 | 17
Not completed — Adverse Event | 9 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Did not take any study medication | 0 | 1
Period: Month 48 Open-Label
Arm/Group | Placebo | Risedronate
Started | 67 | 151
Completed | 55 | 134
Not Completed | 12 | 17
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risedronate | Total
Number analyzed (Participants) | 93 | 192 | 285
Age, Customized [Number; unit: participants] — ITT Population
  participants
    < 65 years | 49 | 120 | 169
    Between 65 and <75 years | 34 | 51 | 85
    >=75 years | 10 | 20 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 93 | 192 | 285
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 7 | 10
  Belgium | 12 | 24 | 36
  Czech Republic | 5 | 12 | 17
  France | 2 | 7 | 9
  United Kingdom | 3 | 6 | 9
  Hungary | 11 | 20 | 31
  Lebanon | 2 | 4 | 6
  Netherlands | 3 | 7 | 10
  Poland | 35 | 73 | 108
  United States | 17 | 32 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), 24 Months/Endpoint, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines. Site will perform at screening to determine if scan should be forwarded to central facility for analysis. Mean of 2 scans performed read by central lab to determine entry qualification. Results standardized (sBMD): Hologic sBMD = 1000 x (BMD x 1.0755), Lunar sBMD = 1000 x (BMD x 0.9522).
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 87 | 188
Percent Change | 1.22 [0.23 to 2.21] | 5.75 [5.00 to 6.50]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; A total of 210 patients will be randomized to 35 mg once a week risedronate and placebo groups in 2:1 ratio. Sample size will allow detection of a difference of at least 3% in lumbar spine BMD percent change from Baseline at 24 months between risedronate and placebo with at least 90% power. This calculation is based on the assumptions that the common within-group standard deviation (SD) would be below 5%, and the dropout rate within 2 years is about 35%; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; Least Square (LS) Mean Difference = 4.53, 95% CI 2-sided [3.46 to 5.60]

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD, Month 6, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines and forwarded to central laboratory for reading.DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines. Results standardized (sBMD): Hologic sBMD = 1000 x (BMD x 1.0755), Lunar sBMD = 1000 x (BMD x 0.9522).
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 86 | 184
Percent Change | 1.03 [0.20 to 1.87] | 3.60 [2.96 to 4.24]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 2.56, 95% CI 2-sided [1.66 to 3.47]

3. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD, Month 12, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines and forwarded to central laboratory for reading. Results standardized (sBMD): Hologic sBMD = 1000 x (BMD x 1.0755), Lunar sBMD = 1000 x (BMD x 0.9522).
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 183
Percent Change | 1.42 [0.51 to 2.34] | 4.60 [3.91 to 5.29]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 3.18, 95% CI 2-sided [2.19 to 4.16]

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD, Month 24, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines and forwarded to central laboratory for reading. Mean of 2 scans performed. Results standardized (sBMD): Hologic sBMD = 1000 x (BMD x 1.0755), Lunar sBMD = 1000 x (BMD x 0.9522).
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 172
Percent Change | 1.40 [0.39 to 2.41] | 5.98 [5.22 to 6.73]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 4.57, 95% CI 2-sided [3.49 to 5.66]

5. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD, Month 6, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines and forwarded to central laboratory for reading. Results standardized (sBMD): Hologic sBMD = 1000 x (1.008 x BMD + 0.006), Lunar sBMD = 1000 x (0.979 x BMD - 0.031).
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 84 | 184
Percent Change | 0.76 [0.22 to 1.31] | 1.16 [0.75 to 1.58]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1856, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 0.40, 95% CI 2-sided [-0.19 to 0.99]

6. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD, Month 12, ITT Population.
Description: as for outcome 5
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 183
Percent Change | 0.74 [0.18 to 1.29] | 1.38 [0.97 to 1.80]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0346, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 0.65, 95% CI 2-sided [0.05 to 1.25]

7. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD, Month 24, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines. Scans will be forwarded to central facility for analysis. Mean of 2 scans performed will be utilized. Results standardized (sBMD): Hologic sBMD = 1000 x (1.008 x BMD + 0.006), Lunar sBMD = 1000 x (0.979 x BMD - 0.031).
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 172
Percent Change | 0.06 [-0.60 to 0.73] | 1.76 [1.26 to 2.26]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 1.70, 95% CI 2-sided [0.98 to 2.41]

8. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD, 24 Months/Endpoint, ITT Population.
Description: as for outcome 7
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 87 | 188
Percent Change | 0.24 [-0.41 to 0.89] | 1.71 [1.21 to 2.20]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 1.46, 95% CI 2-sided [0.76 to 2.17]

9. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Month 6, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines. Scans will be forwarded to central facility for analysis. Baseline femoral neck values measured on Lunar instruments will be normalized to Hologic reference. Hologic Reference BMD = (0.836 x BMD[lunar]) - 0.008
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 84 | 184
Percent Change | 0.48 [-0.32 to 1.27] | 0.98 [0.37 to 1.58]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2538, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 0.50, 95% CI 2-sided [-0.36 to 1.36]

10. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Month 12, ITT Population.
Description: as for outcome 9
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 183
Percent Change | 0.62 [-0.18 to 1.43] | 1.49 [0.88 to 2.10]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0537, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 0.86, 95% CI 2-sided [-0.01 to 1.74]

11. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, Month 24, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines. Scans will be forwarded to central facility for analysis. Mean of 2 scans performed will be utilized. Baseline femoral neck values measured on Lunar instruments will be normalized to Hologic reference. Hologic reference BMD = (0.836 x BMD[lunar]) - 0.008
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 172
Percent Change | 0.42 [-0.43 to 1.27] | 1.65 [1.02 to 2.29]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0081, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 1.24, 95% CI 2-sided [0.32 to 2.15]

12. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD, 24 Months/Endpoint, ITT Population.
Description: as for outcome 11
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 87 | 188
Percent Change | 0.53 [-0.28 to 1.35] | 1.59 [0.97 to 2.21]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0187, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 1.06, 95% CI 2-sided [0.18 to 1.94]

13. Secondary Outcome: Percent Change From Baseline in Femoral Trochanter BMD, Month 6, ITT Population.
Description: DXA (dual energy x-ray absorptiometry) assayed on Lunar or Hologic machines. Scans will be forwarded to central facility for analysis.
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 84 | 184
Percent Change | 0.67 [-0.04 to 1.38] | 1.24 [0.71 to 1.78]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1408, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 0.57, 95% CI 2-sided [-0.19 to 1.34]

14. Secondary Outcome: Percent Change From Baseline in Femoral Trochanter BMD, Month 12, ITT Population.
Description: as for outcome 13
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 183
Percent Change | 0.81 [0.03 to 1.59] | 1.89 [1.30 to 2.48]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0129, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 1.07, 95% CI 2-sided [0.23 to 1.92]

15. Secondary Outcome: Percent Change From Baseline in Femoral Trochanter BMD, Month 24, ITT Population.
Description: as for outcome 13
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 172
Percent Change | 0.52 [-0.37 to 1.41] | 2.83 [2.16 to 3.49]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 2.31, 95% CI 2-sided [1.35 to 3.26]

16. Secondary Outcome: Percent Change From Baseline in Femoral Trochanter BMD, 24 Months/Endpoint, ITT Population.
Description: as for outcome 13
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 87 | 188
Percent Change | 0.57 [-0.29 to 1.44] | 2.73 [2.07 to 3.38]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = 2.15, 95% CI 2-sided [1.22 to 3.08]

17. Secondary Outcome: Percent Change From Baseline in CTx (Type I Collagen C-telopeptide), Month 3, ITT Population.
Time Frame: Baseline to Month 3
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 82 | 180
Percent Change | -14.56 [-21.87 to -7.26] | -58.16 [-63.64 to -52.68]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -43.60, 95% CI 2-sided [-51.52 to -35.67]

18. Secondary Outcome: Percent Change From Baseline in CTx, Month 6, ITT Population.
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 81 | 178
Percent Change | -13.72 [-25.91 to -1.52] | -58.44 [-67.63 to -49.25]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -44.72, 95% CI 2-sided [-58.01 to -31.43]

19. Secondary Outcome: Percent Change From Baseline in CTx, Month 12, ITT Population.
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 175
Percent Change | -19.12 [-31.66 to -6.58] | -61.46 [-70.80 to -52.11]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled centers; LS Mean Difference = -42.33, 95% CI 2-sided [-55.99 to -28.67]

20. Secondary Outcome: Percent Change From Baseline in CTx, Month 24, ITT Population.
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 72 | 163
Percent Change | 9.28 [-2.60 to 21.16] | -37.27 [-46.06 to -28.48]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -46.55, 95% CI 2-sided [-59.38 to -33.72]

21. Secondary Outcome: Percent Change From Baseline in CTx, 24 Months/Endpoint, ITT Population.
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 183
Percent Change | 6.39 [-4.55 to 17.34] | -38.76 [-46.97 to -30.54]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -45.15, 95% CI 2-sided [-57.01 to -33.29]

22. Secondary Outcome: Percent Change From Baseline in NTx/Cr (Type I Collagen N-telopeptide/Creatinine), Month 3, ITT Population.
Time Frame: Baseline to Month 3
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 84 | 181
Percent Change | -17.41 [-24.38 to -10.43] | -33.28 [-38.58 to -27.98]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -15.88, 95% CI 2-sided [-23.43 to -8.32]

23. Secondary Outcome: Percent Change From Baseline in NTx/Cr, Month 6, ITT Population.
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 180
Percent Change | -7.98 [-16.33 to 0.38] | -29.97 [-36.34 to -23.60]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -22.00, 95% CI 2-sided [-31.08 to -12.91]

24. Secondary Outcome: Percent Change From Baseline in NTx/Cr, Month 12, ITT Population.
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 176
Percent Change | -16.46 [-24.55 to -8.37] | -38.42 [-44.45 to -32.39]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -21.96, 95% CI 2-sided [-30.75 to -13.17]

25. Secondary Outcome: Percent Change From Baseline in NTx/Cr, Month 24, ITT Population.
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 75 | 167
Percent Change | -22.27 [-30.69 to -13.85] | -37.38 [-43.69 to -31.07]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0012, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -15.11, 95% CI 2-sided [-24.20 to -6.02]

26. Secondary Outcome: Percent Change From Baseline in NTx/Cr, 24 Months/Endpoint, ITT Population.
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 85 | 186
Percent Change | -20.45 [-28.68 to -12.23] | -36.82 [-43.04 to -30.60]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -16.37, 95% CI 2-sided [-25.24 to -7.49]

27. Secondary Outcome: Percent Change From Baseline in BAP (Bone-specific Alkaline Phosphatase), Month 3, ITT Population.
Time Frame: Baseline to Month 3
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 82 | 179
percent | -8.89 [-12.25 to -5.53] | -24.53 [-27.05 to -22.00]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -15.64, 95% CI 2-sided [-19.29 to -11.99]

28. Secondary Outcome: Percent Change From Baseline in BAP, Month 6, ITT Population.
Time Frame: Baseline to Month 6
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 81 | 178
Percent Change | -8.68 [-12.82 to -4.54] | -29.78 [-32.90 to -26.66]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -21.10, 95% CI 2-sided [-25.61 to -16.59]

29. Secondary Outcome: Percent Change From Baseline in BAP, Month 12, ITT Population.
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 175
Percent Change | -7.11 [-12.08 to -2.14] | -29.51 [-33.21 to -25.81]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -22.39, 95% CI 2-sided [-27.80 to -16.98]

30. Secondary Outcome: Percent Change From Baseline in BAP, Month 24, ITT Population.
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 72 | 163
percent | 2.95 [-7.87 to 13.77] | -25.20 [-33.20 to -17.20]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -28.15, 95% CI 2-sided [-39.84 to -16.47]

31. Secondary Outcome: Percent Change From Baseline in BAP, 24 Months/Endpoint, ITT Population.
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 83 | 183
Percent Change | 1.99 [-7.60 to 11.57] | -25.27 [-32.46 to -18.07]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -27.25, 95% CI 2-sided [-37.63 to -16.87]

32. Secondary Outcome: Change From Baseline in Body Height, Month 12, ITT Population.
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 82 | 183
millimeters | -0.77 [-2.49 to 0.94] | -0.92 [-2.20 to 0.37]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8794, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -0.14, 95% CI 2-sided [-1.99 to 1.71]

33. Secondary Outcome: Change From Baseline in Body Height, Month 24, ITT Population.
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 176
millimeters | -2.66 [-4.67 to -0.65] | -3.13 [-4.62 to -1.64]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6658, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -0.47, 95% CI 2-sided [-2.62 to 1.67]

34. Secondary Outcome: Change From Baseline in Body Height, 24 Months/Endpoint, ITT Population.
Time Frame: Baseline to 24 Months/Endpoint
Population: ITT Population, LOCF (Last Observation Carried Forward)
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 84 | 189
millimeters | -2.39 [-4.34 to -0.44] | -2.68 [-4.14 to -1.22]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7840, ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -0.29, 95% CI 2-sided [-2.39 to 1.81]

35. Secondary Outcome: Percent of Responders Lumbar Spine BMD, Month 24, ITT Population
Description: responder = positive change (>0) in lumbar spine BMD from Baseline to Month 24
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 78 | 172
Percentage of Participants | 60.3 | 89.5
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Controlled for pooled center

36. Secondary Outcome: Cumulative Incidence of Fractures, 12 Months, ITT Population
Description: Kaplan-Meier Cumulative Incidence, fractures / 100 patients / year
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Number; unit: Fractures / 100 patients / year
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 92 | 191
Fractures / 100 patients / year | 3.4 | 2.7
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7284, Log Rank; Relative Risk = 0.771, 95% CI [0.184 to 3.226]

37. Secondary Outcome: Cumulative Incidence of Fractures, 24 Months, ITT Population
Description: Kaplan-Meier Cumulative Incidence, fractures / 100 patients / 2 years
Time Frame: Baseline to Month 24
Population: ITT Population
Measure: Number; unit: Fractures / 100 patients / 2 years
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 92 | 191
Fractures / 100 patients / 2 years | 7.7 | 4.9
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5293, Log Rank; Relative Risk = 0.688, 95% CI 2-sided [0.245 to 1.932]

ADVERSE EVENTS:
Time Frame: 2 year double-blind treatment followed by 2 year open-label treatment.
Description: Year 2, 93 placebo and 191 Risedronate patients with Most Frequent AE threshold of 3%. Year 4, 67 placebo to Risedronate patients and 151 Risedronate/Risedronate patients with Most Frequent AE threshold of 2%.
Groups:
- Placebo Year 2: Placebo tablet once weekly Years 1 & 2
- Risedronate Year 2: Risedronate 35 mg tablet once weekly Years 1 & 2
- Placebo-Risedronate Year 4: Placebo once weekly Years 1 & 2 followed by risedronate 35 mg once weekly Years 3 & 4
- Risedronate Year 4: Risedronate 35 mg tablet once weekly Years 1 thru 4
Arm/Group | Placebo Year 2 | Risedronate Year 2 | Placebo-Risedronate Year 4 | Risedronate Year 4
Serious Adverse Events (participants affected / at risk) | 15/93 | 29/191 | 8/67 | 21/151
Other Adverse Events (participants affected / at risk) | 66/93 | 134/191 | 46/67 | 97/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Year 2 (N=93) | Risedronate Year 2 (N=191) | Placebo-Risedronate Year 4 (N=67) | Risedronate Year 4 (N=151)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteritis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atherosclerosis Obliterans (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchioloalveolar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis Acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burns Third Degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastritis Atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 3 (5) | 1 (1) | 1 (1) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Prostate Examination Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Cell Lung Cancer, Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden Cardiac Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Year 2 (N=93) | Risedronate Year 2 (N=191) | Placebo-Risedronate Year 4 (N=67) | Risedronate Year 4 (N=151)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (13) | 2 (2) | 7 (8)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 4 (5) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 13 (14) | 3 (3) | 10 (12)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 3 (3) | 9 (9) | 3 (3) | 5 (5)
Chest Pain (General disorders) | 4 (4) | 4 (5) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 16 (17) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 5 (6) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 10 (10) | 0 (0) | 9 (9)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 5 (5) | 1 (1) | 11 (11)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 11 (11) | 1 (1) | 4 (4)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 11 (13) | 2 (2) | 12 (15)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (9) | 0 (0) | 5 (5)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Prostate Examination Abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 7 (8) | 2 (2) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less